CLINICAL TRIAL: NCT04193501
Title: Frequency of Sleep Abnormalities in Patients With Irritable Bowel Syndrome and Its Relationship With Symptom Severity, Quality of Life and Effect of Pharmacological Intervention to Improve Sleep on These Parameters
Brief Title: Frequency of Sleep Abnormalities in Patients With Irritable Bowel Syndrome and Effect of Pharmacological Intervention
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2018-207-EMP-107
Record Dates: First submitted 2019-10-28; First posted 2019-12-10 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2019-12

CONDITIONS: Irritable Bowel Syndrome
Keywords: Melatonin; gut microbiota; dysbiosis
MeSH Terms: conditions — Irritable Bowel Syndrome; Dysbiosis | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: Randomized, Parallel Group, Placebo Controlled Trial
Who Masked: Participant, Investigator
Masking Description: Participant and Investigator Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arms (Experimental): Melatonin dose: 3mg/OD
  Interventions: Drug: Melatonin 3 mg
- Control arms (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Melatonin 3 mg — Melatonin dose: 3mg/OD Melatonin is a hormone made by the pineal gland; its biosynthesis is initiated by the uptake of the essential amino acid tryptophan and is an important inducer of sleep. Abnormality in melatonin has been shown in several studies on patients of IBS and functional constipation.
  Other Names: 5-Methoxy-N-Acetyltryptamine
  Arms: Experimental arms
Other: Placebo — Similar looking placebo
  Arms: Control arms

SUMMARY:
Irritable bowel syndrome (IBS), a common gastrointestinal (GI) disorder in India and in the rest of the World, is enigmatic in its pathogenesis. IBS is associated with recurrent abdominal pain or discomfort, bloating, incomplete evacuation, altered bowel habits, and abnormal stool forms. The etiology of IBS remains unclear and different factors were thought to be involved like genetics and environmental factors, visceral hypersensitivity, altered gut microbiota or disorder of the microbiota-gut-brain axis and various psychological factors like anxiety, depression, and insomnia or sleep disturbance. Due to increasing work pressure in today's society, and the consequent shift duty and psychological stress, the frequency of sleep disorders is increasing; disturbed sleep may be associated with a vicious cycle in which altered sleep may result in gastrointestinal (GI) disturbances, which in turn, may jeopardize sleep further. The disorder of the gut microbiota, the largest organ of the human body, is being suggested to be responsible for several GI and extra-GI diseases. Qualitative change in gut microbiota is currently studied by next-generation sequencing. Gut and sleep patterns work in an axis - a two-way street of communication, some studies reported altered gut microbiota or dysbiosis modulates peripheral and central nervous system function, leading to alterations in brain signaling and behavior that possibly leads to sleep disturbances.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS), a common gastrointestinal (GI) disorder in India and in the rest of the World, is enigmatic in its pathogenesis. IBS is associated with recurrent abdominal pain or discomfort, bloating, incomplete evacuation, altered bowel habits, and abnormal stool forms. The etiology of IBS remains unclear and different factors were thought to be involved like genetics and environmental factors, visceral hypersensitivity, altered gut microbiota or disorder of the microbiota-gut-brain axis and various psychological factors like anxiety, depression, and insomnia or sleep disturbance. Due to increasing work pressure in today's society, and the consequent shift duty and psychological stress, the frequency of sleep disorders is increasing; disturbed sleep may be associated with a vicious cycle in which altered sleep may result in gastrointestinal (GI) disturbances, which in turn, may jeopardize sleep further. The disorder of the gut microbiota, the largest organ of the human body, is being suggested to be responsible for several GI and extra-GI diseases. Qualitative change in gut microbiota is currently studied by next-generation sequencing. Gut and sleep patterns work in an axis - a two-way street of communication, some studies reported altered gut microbiota or dysbiosis modulates peripheral and central nervous system function, leading to alterations in brain signaling and behavior that possibly leads to sleep disturbances.

Several case-control and meta-analyses have reported an association between sleep disturbance and irritable bowel syndrome (IBS) as compared to healthy controls. However, the data regarding the relationship between sleep disturbance and severity parameters of IBS have not been widely reported; moreover, interventions that improve disturbed sleep on these parameters are scanty. There is no systematic study on sleep disorders among patients with IBS from India.

Melatonin is a hormone made by the pineal gland; its biosynthesis is initiated by the uptake of the essential amino acid tryptophan and is an important inducer of sleep. Abnormality in melatonin has been shown in several studies on patients of IBS and functional constipation. A few studies also reported improvement in sleep and GI function after the administration of melatonin. However, these studies had limitations due to the small sample size, lack of randomization and inclusion of patients without the sleep disorder. Moreover, there is no study from India on this issue.

Accordingly, investigators wish to undertake a study with the following aims: (i) Quality of sleep among patients with IBS and healthy controls. (ii) Levels of 6-Hydroxymelatonin sulphate (a metabolite of melatonin) both in patients with IBS and healthy controls.

(iii) Relationship between the IBS symptom severity (IBS-SSS), Health-Related Quality of Life (HRQL) and sleep disorder and melatonin deficiency, (iv) Relationship between sleep quality and rectal sensory function (by barostat) (v) Relationship between gut dysbiosis and the IBS symptom severity (IBS-SSS), Health-Related Quality of Life (HRQL) and sleep disorder (vi) Effect of melatonin administration on IBS symptoms, HRQL, and sleep. Since sleep disturbance may be an important issue in IBS, the patients with IBS will be treated both with melatonin and standard treatment. Parameters like IBS-SSS, HRQL, Hospital Anxiety and Depression Scale (HADS) score, Pittsburgh Sleep Quality Index (PSQI) will be studied in patients with IBS and healthy controls and these parameters would be repeated after 1 and 3 months follow-up in patients only. Urinary 6-Hydroxymelatonin sulphate will be studied in patients and controls before treatment with standard medical therapy (SMT) plus melatonin and it will be repeated after one month among patients with IBS only. The sleep study will be performed by the PSQI questionnaire and also by polysomnography depending on the availability of the instrument. The rectal sensory function will be studied by barostat. The study will analyse the effect of melatonin in GI and sleep disorder functions. Data will be analyzed using appropriate statistical techniques. P-values lesser than 0.05 will be considered significant.

Study protocol:

Sample size:

The related case-control studies were reviewed for the calculation of sample size. The frequency of sleep disorder among IBS was observed to be 35% and 43% whereas in control it has been observed to be 29 and 14% respectively. Taking the average of these, investigators considered among IBS case and controls the average frequency of sleep disorder is 40% and 22%, respectively, considering a power of 80%, alpha value of 0.05 and ratio of the case to control is 1:1. As per the calculation, investigators propose to include 97 cases and 97 controls.

For an interventional study with SMT plus melatonin and SMT plus placebo, the sample size was calculated based on the data that improvement occurred in 88% patients if treated with SMT plus melatonin as compared to 47% with SMT plus placebo. Hence, 34 patients will be treated with SMT plus melatonin and 34 with SMT plus placebo (two-sided CI 99%, power 80%, case: control 1:1, and p-value <0.05). Considering 20-25% loss to follow-up, 97 patients with IBS will be randomized to SMT plus melatonin and SMT plus placebo.

Actual plan of work:

Study site:

This study will be conducted in the Department of Gastroenterology, in inter-departmental collaborations with the Department of Neurology to analyse the effect of SMT plus melatonin in GI and sleep.

Inclusion criteria

* Diagnosis by ROME III/IV criteria.
* Willing to participate and informed consent is obtained. Exclusion criteria
* Presence of alarm symptoms such as severe organic GI diseases, unexplained iron deficiency anaemia, unintentional weight loss, palpable abdominal mass.
* No active substance intake.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis by ROME III/IV criteria.
* Willing to participate and informed consent is obtained.

Exclusion Criteria:

* Presence of alarm symptoms such as severe organic GI diseases, unexplained iron deficiency anemia, unintentional weight loss, palpable abdominal mass.
* No active substance intake.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Change in levels of 6-Hydroxymelatonin sulphate | 1 month
  To study changes from baseline, in levels of 6-Hydroxymelatonin sulphate (a metabolite of melatonin) both in patients with IBS and healthy controls
Sleep quality index score | 1 month
  Self-reported usual sleep habits for the majority of days and nights during the past month only. The 19 self-rated and 5 non-self rated questions combined to form seven component scores, with a range of 0-21 points, "0" indicating no difficulty and "21" indicating severe difficulties.

SECONDARY OUTCOMES:
Change in IBS symptom severity scores | 1 month and 3 months
  Remission or response (patients scoring between 75-175 and controls below 75) after 1 month and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Uday C Ghoshal, Principal Investigator — Medical council of India, Association of Indian Universities
Locations (2):
- India (2):
  - Department of Critical Care Medicine, SGPGIMS, Lucknow, Uttar Pradesh
  - Sanjay Gandhi Postgraduate Institute of Medical Sciences (SGPGIMS), Lucknow, Uttar Pradesh

IPD SHARING:
Plan to Share IPD: No
This study will be conducted in the Department of Gastroenterology, in inter-departmental collaborations with the department of Neurology to analyse the effect of SMT plus melatonin in GI and sleep.

REFERENCES:
- [Result] Ghoshal UC, Shukla A. Malnutrition in inflammatory bowel disease patients in northern India: frequency and factors influencing its development. Trop Gastroenterol. 2008 Apr-Jun;29(2):95-7. PMID 18972769

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/01/NCT04193501/Prot_ICF_000.pdf